CLINICAL TRIAL: NCT05961852
Title: COmbiNing Cutting and Drug-Eluting Balloon for Resistant Arteriovenous Fistula sTenOsis (CONCERTO)
Acronym: CONCERTO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONCERTO
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Arteriovenous Fistula Stenosis
Keywords: arteriovenous fistula; drug-coated balloon; cutting balloon; stenosis
MeSH Terms: conditions — Arteriovenous Fistula; Constriction, Pathologic | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Cutting and drug-coated balloon angioplasty
  Interventions: Device: Angioplasty

INTERVENTIONS:
Device: Angioplasty — Angioplasty with cutting and drug-coated balloon

SUMMARY:
To evaluate the preliminary efficacy of combination of cutting and drug-coated balloon for the treatment of resistant AVF stenosis.

DETAILED DESCRIPTION:
This is a single arm pilot study recruiting 19 participants with resistant AVF stenosis (defined as having > 30% residual stenosis after optimal balloon angioplasty) to receive cutting and drug-coated balloon.

The outcome measure is target lesion primary patency at 6 months. Outcome will be clinically driven.

ELIGIBILITY:
Inclusion Criteria:

1. Failing mature upper limb AVF
2. Resistant stenosis (>30% residual stenosis) after optimal conventional balloon angioplasty (appropriately sized balloon, inflated up to rated burst pressure, at least twice for at least a minute per inflation)
3. Patient is >= 21 years of age
4. Ability to provide informed consent

Exclusion Criteria:

1. Thrombosed AVF
2. Target lesion has a sharp angle (> 45 degrees)
3. Lesions requiring cutting balloon size > 7 mm
4. Coagulopathy or thrombocytopaenia that cannot be adequately managed for the procedure
5. Contraindication to dual antiplatelet therapy
6. Severe allergy to contrast media that cannot be adequately managed for the procedure
7. Breast-feeding and/or pregnant females
8. Male patients who are planning to father children during the trial period
9. Unable to comply with follow up protocol (for instance, limited life expectancy)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Target lesion primary patency | 6 months after index procedure
  Time from index treatment to repeat treatment of target lesion or thrombosis of circuit.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Da Zhuang, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu CC, Lin MC, Pu SY, Tsai KC, Wen SC. Comparison of cutting balloon versus high-pressure balloon angioplasty for resistant venous stenoses of native hemodialysis fistulas. J Vasc Interv Radiol. 2008 Jun;19(6):877-83. doi: 10.1016/j.jvir.2008.02.016. Epub 2008 May 2. PMID 18503902